CLINICAL TRIAL: NCT05501314
Title: Remote Home Monitoring of Patients With a Predicted Mild Acute Pancreatitis - A Feasibility Study (REMAP)
Brief Title: Remote Home Monitoring Acute Pancreatitis
Acronym: REMAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rijnstate Hospital (Other)
Collaborators: University of Twente (Other); Philips Research Eindhoven (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NL81630.091.22
Record Dates: First submitted 2022-08-08; First posted 2022-08-15 (Actual); Last update posted 2022-08-15 (Actual); Status verified 2022-08

CONDITIONS: Acute Pancreatitis; Telemedicine; Healthdot; Patient Discharge; Monitoring
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Intervention Model Description: Feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Early discharge with remote home monitoring. (Experimental): * Patients are discharged early
  * Patients receive remote home monitoring using a wearable sensor and a smartphone app.
  * Patients fill in a satisfaction questionnaire
  Interventions: Other: Early discharge with remote home monitoring.

INTERVENTIONS:
Other: Early discharge with remote home monitoring. — After at least 48 hours of hospital admission, patients are discharged early with the use of remote home monitoring. During home monitoring, heartrate, respiratory rate, posture and movement are monitored every 5 minutes for at least 4 days, using a wearable sensor. Core temperature is monitored using an ear thermometer. Patients are contacted once per day by a nurse from the Virtual Monitoring Centre (VMC) to assess pancreatitis related complaints, intake of fluids and food, pain and the use of analgesics. Patients are asked to provide information to the hospital using a smartphone app.

SUMMARY:
Acute pancreatitis is an inflammation of the pancreas which causes abdominal pain and is the most common gastro-intestinal reason for acute hospitalization in Western countries. Because care for a mild acute pancreatitis is supportive, early discharge of patients with a predicted mild course of acute pancreatitis might be safe with the use of remote home monitoring. This might reduce the demand for hospital beds and allow patients to benefit from recovering in their home environment. Therefore, the aim of this study is to assess the feasibility of a novel care pathway in which patients with a predicted mild course of acute pancreatitis are discharged early with remote home monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Have 2 out of 3 revised Atlanta criteria for pancreatitis:

  * Abdominal pain consistent with acute pancreatitis
  * Serum lipase ≥ 3x upper limit normal (> 159 U/l)
  * Typical pancreatic abnormalities on imaging (ultrasound, CT or MRI)
* First episode of acute pancreatitis or a prior pancreatitis more than 3 months ago.
* Age ≥18 years, both men and women.
* Able and willing to provide written informed consent.
* In possession of a working (smart)phone on which patient can be reached for the duration of participation (30 days).

Exclusion Criteria:

* Chronic pancreatitis according to M-ANNHEIM criteria (20).
* Signs of severe pancreatitis at the moment of admission to the GE ward:

  * Serum CRP > 150 mg/l
  * More than one SIRS criteria:

    * temperature < 36◦C or > 38◦C
    * heart rate > 90/min
    * respiratory rate >20/min
    * leucocytes < 4x/109l or > 12x109/l
* MEWS (Modified Early Warning Score) ≥6 or in need of ICU admission
* Living alone or in an institution (e.g. psychiatric ward or nursing home)
* Known sensitivity to medical adhesives
* Known pregnancy
* Have one or more of the following comorbidities:

  * Heart failure (NYHA class III or IV)
  * COPD (Gold III-IV)
  * Kidney disease (>G3b) and/or kidney replacement therapy
  * Currently undergoing oncological treatment
  * Use of immunosuppressants
  * Dysregulated or poorly controlled insulin dependent diabetes
  * Morbid obesity (BMI>35 kg/m2)
  * Implantable Cardioverter Defibrillator (ICD) or Pacemaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Incidence (%) of unplanned hospital readmissions. | Within 30 days of discharge
  To determine the feasibility of novel care pathway
2. Incidence (%) of pancreatitis related complications. These complications include necrotizing pancreatitis, infection, pseudocysts, new onset diabetes, recurrence of pancreatitis, cholecystitis or cholangitis. | Within 30 days of discharge
  To determine the feasibility of novel care pathway
3. Mortality (%) of patients discharged home with remote monitoring. | Within 30 days of discharge
  To determine the feasibility of novel care pathway

SECONDARY OUTCOMES:
Length of stay in the hospital | Within 30 days of discharge.
The amount of extra contacts between VMC-nurse or physician and the patient, in addition to the usual call once per day as documented in the smartphone app. | Within 30 days of discharge
The amount of laboratory or imaging tests | Within 30 days of discharge
  All bloodtests and imaging tests (US, MRI and CT-scan will be documented)
Amount of adjustments in analgesics needed during home monitoring | Within 30 days of discharge

OTHER OUTCOMES:
Patient satisfaction is assessed using a satisfaction questionnaire | After 14 days of discharge.
  Using a combination of two validated questionnaires
Overall costs of treatment | Within 30 days of discharge

CONTACTS AND LOCATIONS:
Overall Officials: C.M.J. Doggen, prof. dr., Principal Investigator — Rijnstate Hospital
Locations (1):
- Rijnstate Hospital, Arnhem, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes